CLINICAL TRIAL: NCT05944419
Title: Influence of Neck Design on Peri-implant Hard and Soft Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jordi caballé, Dr, MSc, PhD, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIR-ECL-2016-05
Record Dates: First submitted 2023-06-07; First posted 2023-07-13 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Bone Resorption; Soft Tissue Bleeding
Keywords: dental implants; implant neck design; immediate implants; immediate provisionalization; buccal bone thickness
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- V3 Implant MIS Iberica (Active Comparator): Implant with triangular neck macro design
  Interventions: Device: Immediate implant surgery
- C1 Implant MIS Iberica (Active Comparator): Implant with circular neck macro design
  Interventions: Device: Immediate implant surgery

INTERVENTIONS:
Device: Immediate implant surgery — Placement of immediate implant and immediate provisionalization after tooth extraction

SUMMARY:
The goal of this clinical trial is to test two different implant neck designs in 36 patients. The main question[s] it aims to answer are:

* do triangular neck designed implants placed immediately after dental extraction have the same influence on peri-implant hard and soft tissues than regular neck designed implants at one year?
* do triangular neck designed implants placed immediately after dental extraction have the same influence on peri-implant hard and soft tissues than regular neck designed implants at three years?

Participants that present an unrepairable tooth on the anterior upper maxilla will be asked to take a CBCT scan in order to verify the presence of the buccal bone. Once this is verified the patients will enter in the study and the day of the surgery they will be assigned to either control or test group.

* Control group: C1 round-neck implant
* Test groups: V3 triangular-implant neck

Researchers will compare test and control groups to see if they have the same effects on hard and soft tissues at 4 months, 1 year and 3 years.

DETAILED DESCRIPTION:
Immediate implant placement is considered to be a technique-sensitive protocol with a variety of potential risks. The interface area between the neck of the implant and the abutment is critical; it can affect the treatment outcome, particularly mar-ginal bone loss (MBL) and soft tissue behavior. Traditionally, the implant neck is circu-lar in shape; however, a new triangular neck design has recently been introduced on the market, though advanced indications of this innovative design are still lacking.

The objective of this randomized clinical trial was to compare the clinical and radiographic outcomes obtained after immediate placement of implants and temporization of two different neck geometries: a traditional round neck (RN) and an innovative neck with a triangular shape (TN).

ELIGIBILITY:
Inclusion Criteria:

* healthy non-smokers or light smokers (< 10 cigarettes/day)
* adults (> 18 years of age),
* need for single tooth extraction of a maxillary incisor, canine or premolar
* adequate oral hygiene
* ability to follow instructions and attend the required appointments
* presence of a length of at least 3 mm of buccal bone measuring ≥ 0.5 mm in thickness, apical to the extraction socket
* stable and intact socket walls

Exclusion Criteria:

* patients with acute infections in the area of interest
* individuals with large occlusal discrepancies and/or occlusal overload para-functions
* smokers of more than 10 cigarettes/day
* patients with any medical condition or medication contraindicating dental implant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Buccal bone width (BBW) | 4 months
  buccal bone width was measured by CBCT (iCAT®, Imaging Science International, LLC, Hatfield, PA, USA) at four points: at the implant neck, and at 1 mm, 2 mm and 3 mm above the implant neck.
Marginal bone loss (MBL) | 4 months
  marginal bone loss was measured on mesial and distal aspects of the implant using intraoral standardized periapical radiographs with the parallel technique. Measurements were performed using K-Pacs Work-station (Image Information Systems, Ltd.). The distance from the implant shoulder to the first bone-implant contact was measured at the mesial and distal sites.
Marginal bone loss (MBL) | 1 years
  marginal bone loss was measured on mesial and distal aspects of the implant using intraoral standardized periapical radiographs with the parallel technique. Measurements were performed using K-Pacs Work-station (Image Information Systems, Ltd.). The distance from the implant shoulder to the first bone-implant contact was measured at the mesial and distal sites.
Marginal bone loss (MBL) | 3 years
  marginal bone loss was measured on mesial and distal aspects of the implant using intraoral standardized periapical radiographs with the parallel technique. Measurements were performed using K-Pacs Work-station (Image Information Systems, Ltd.). The distance from the implant shoulder to the first bone-implant contact was measured at the mesial and distal sites.
Soft tissue thickness (STT) | 4 months
  the thickness of the buccal soft tissue at 3 mm and 5 mm from the gingi-val margin was measured using an endodontic file.
Soft tissue thickness (STT) | 1 years
  the thickness of the buccal soft tissue at 3 mm and 5 mm from the gingi-val margin was measured using an endodontic file.
Soft tissue thickness (STT) | 3 years
  the thickness of the buccal soft tissue at 3 mm and 5 mm from the gingi-val margin was measured using an endodontic file.

SECONDARY OUTCOMES:
Insertion torque (IT): | day 1
  the insertion torque of the implant was measured on the day of the sur-gery with the implant motor.
ISQ (implant stability quotient): | day 1
  the ISQ was measured at implant placement using the Osstell device, which involves resonance frequency analysis (RFA) for measuring the fre-quency of vibration.
Probing pocket depth (PPD): | 4 months
  probing pocket depth was measured with a Marquis Color code dental probe at 6 sites covering 360ª of the tooth: three on the buccal site and three on the palatal site of each tooth.
Probing pocket depth (PPD): | 1 year
  probing pocket depth was measured with a Marquis Color code dental probe at 6 sites covering 360ª of the tooth: three on the buccal site and three on the palatal site of each tooth.
Probing pocket depth (PPD): | 3 year
  probing pocket depth was measured with a Marquis Color code dental probe at 6 sites covering 360ª of the tooth: three on the buccal site and three on the palatal site of each tooth.
Bleeding on probing (BOP): | 4 months
  bleeding on probing was registered at each PPD site, whether there was bleeding or not.
Bleeding on probing (BOP): | 1 year
  bleeding on probing was registered at each PPD site, whether there was bleeding or not.
Bleeding on probing (BOP): | 3 year
  bleeding on probing was registered at each PPD site, whether there was bleeding or not.
Crestal width (CW) | 4 months
  at 3 mm and 5 mm from the gingival margin: a gauge compass was used to measure the whole width of the crestal volume, from palatal to ves-tibular wall.
Crestal width (CW) | 1 year
  at 3 mm and 5 mm from the gingival margin: a gauge compass was used to measure the whole width of the crestal volume, from palatal to ves-tibular wall.
Crestal width (CW) | 3 year
  at 3 mm and 5 mm from the gingival margin: a gauge compass was used to measure the whole width of the crestal volume, from palatal to ves-tibular wall.
Pink esthetic score (PES): | 4 months
  this score was measured based on the Furhauser table. Maximum: 14 points / Minimum: 0 points. Higher scores mean a better outcome.
Pink esthetic score (PES): | 1 year
  this score was measured based on the Furhauser table. Maximum: 14 points / Minimum: 0 points. Higher scores mean a better outcome.
Pink esthetic score (PES): | 3 year
  this score was measured based on the Furhauser table. Maximum: 14 points / Minimum: 0 points. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: CRISTINA PORTA FERRER, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- [Derived] Porta-Ferrer C, Elnayef-Elsakan B, Del Amo FS, Caballe-Serrano J, Satorres-Nieto M, Hernandez-Alfaro F. Influence of Neck Design on Peri-Implant Hard and Soft Tissues: A 12-Month Randomized Clinical Trial of Immediately Placed Implants. Clin Oral Implants Res. 2025 Nov 23. doi: 10.1111/clr.70068. Online ahead of print. PMID 41275475